CLINICAL TRIAL: NCT02102763
Title: Greek Childhood Obesity Study
Brief Title: Greek Childhood Obesity (GRECO) Study
Acronym: GRECO
Status: Completed | Type: Observational
Sponsor: Agricultural University of Athens (Other)
Collaborators: General Secretariat of Consumers-Greek Ministry of Development (Unknown); Hellenic Association of Food and Beverage Companies (Unknown); Coca Cola Hellas (Unknown); Coca Cola Hellenic Bottling Company (Unknown); Cereal Partners Hellas (Unknown); FAGE S.A. (Unknown); Unilever Hellas (Unknown); Nestle Hellas (Unknown); Kraft Foods Hellas (Unknown); European Union and Greek national funds - Research Funding Program: Heraclitus II. (Unknown)
Responsible Party: Principal Investigator, Paul Farajian, Dr Paul Farajian, Agricultural University of Athens
Other Study IDs: AgriculturalUA
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Overweight; Obesity; Dietary Habits; Physical Activity; Blood Pressure
Keywords: Overweight; Obesity; Dietary intake; Physical activity levels; Blood pressure levels; Family perceptions
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the GRECO study were to: a) to provide national data on overweight and obesity prevalence in a representative sample of primary schoolchildren aged 10-12 years old, b) to identify those socio-economic, demographic factors, as well as dietary and physical activity habits and familial characteristics that are associated with childhood and preadolescent overweight and obesity, c) to identify lifestyle and dietary patterns that are associated with elevated blood pressure levels and dietary sodium intake.

ELIGIBILITY:
Inclusion Criteria:

* Within the age range
* 5th and 6th grade public schools children
* Consent form provided by the parents

Exclusion Criteria:

* Not providing signed parental consent forms
* Outside the required age range

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A nationwide cross-sectional sample of 10-12 years old Greek schoolchildren
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Overweight and obesity prevalence in a representative sample of primary schoolchildren aged 10-12 years old | 8 months
  Assessment of overweight and obesity by measuring body weight and standing height. Body mass index was calculated by dividing weight (kg) by standing height squared (m2). Obesity and overweight among children were calculated using the International Obesity Task Force (IOTF) age and gender specific body mass index cut-off criteria

SECONDARY OUTCOMES:
Dietary intake assessment | 8 months
  Dietary assessment was based on a validated self-reported, semi-quantitative picture-aid food frequency questionnaire (FFQ), consisted of 48 food items commonly used in the local Greek cuisine.
Assessment of eating behaviors | 8 months
  Assessment of the frequency of breakfast consumption and number of eating occasions (number of meals and snacks during the day), as well as the frequency of having meals in front of a screen (watching television/DVD/videos and/or using of games consoles/computer), and the frequency of having meals together with the whole family or at least with one family member.
Assessment of physical activity and inactivity levels | 8 months
  Physical activity levels assessment was performed by the Physical Activity Questionnaire for older Children. Children were also asked whether they had television or computer in their room and were asked to report the average weekdays and weekend time (h/d) spent on sedentary activities and more specifically on watching television/DVD/movies and/or recreational usage of games consoles/computer.

OTHER OUTCOMES:
Blood pressure measurements | 8 months
  Blood pressure was measured in a single occasion within the schools' settings using validated oscillometric devices

CONTACTS AND LOCATIONS:
Overall Officials: Paul Farajian, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Department of Food Science and Human Nutrition, Agricultural University of Athens, Athens, Attica, Greece

REFERENCES:
- [Background] Farajian P, Risvas G, Karasouli K, Pounis GD, Kastorini CM, Panagiotakos DB, Zampelas A. Very high childhood obesity prevalence and low adherence rates to the Mediterranean diet in Greek children: the GRECO study. Atherosclerosis. 2011 Aug;217(2):525-30. doi: 10.1016/j.atherosclerosis.2011.04.003. Epub 2011 Apr 13. PMID 21561621
- [Background] Magriplis E, Farajian P, Pounis GD, Risvas G, Panagiotakos DB, Zampelas A. High sodium intake of children through 'hidden' food sources and its association with the Mediterranean diet: the GRECO study. J Hypertens. 2011 Jun;29(6):1069-76. doi: 10.1097/HJH.0b013e328345ef35. PMID 21451420
- [Background] Farajian P, Panagiotakos DB, Risvas G, Karasouli K, Bountziouka V, Voutzourakis N, Zampelas A. Socio-economic and demographic determinants of childhood obesity prevalence in Greece: the GRECO (Greek Childhood Obesity) study. Public Health Nutr. 2013 Feb;16(2):240-7. doi: 10.1017/S1368980012002625. Epub 2012 May 25. PMID 22625663
- [Background] Risvas G, Papaioannou I, Panagiotakos DB, Farajian P, Bountziouka V, Zampelas A. Perinatal and family factors associated with preadolescence overweight/obesity in Greece: the GRECO study. J Epidemiol Glob Health. 2012 Sep;2(3):145-53. doi: 10.1016/j.jegh.2012.06.002. Epub 2012 Aug 18. PMID 23856452